CLINICAL TRIAL: NCT02256800
Title: Determination of the UGT1A1 Polymorphism as Guidance for Irinotecan Dose Escalation in Metastatic Colorectal Cancer Treated With First-Line Bevacizumab and FOLFIRI (PURE FIST)
Brief Title: Escalated Dose of Irinotecan in mCRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaw-Yuan Wang, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Jaw-Yuan Wang, MD, PhD, Professor, Kaohsiung Medical University Chung-Ho Memorial Hospital
Organization: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-20130020
Record Dates: First submitted 2014-09-18; First posted 2014-10-06 (Estimated); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — UGT1A1 enzyme; Bevacizumab; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- UGT1A1 genotyping (6,6) (Experimental): The investigators will escalate the dosage of irinotecan from 180mg/m2 to 260 mg/m2
  Interventions: Genetic: UGT1A1 genotyping (6,6); Drug: bevacizumab (Avastin); Drug: irinotecan; Drug: Leucovorin; Drug: 5-FU
- UGTA1T1 genotyping (6,7) (Experimental): The investigators will escalate the dosage of irinotecan from 180mg/m2 to 240 mg/m2
  Interventions: Genetic: UGTIA1 genotyping (6,7); Drug: bevacizumab (Avastin); Drug: irinotecan; Drug: Leucovorin; Drug: 5-FU
- UGTA1T1 genotyping (7,7) (Experimental): The investigators will escalate the dosage of irinotecan from 120mg/m2 to 180 mg/m2
  Interventions: Genetic: UGTIA1 genotyping (7,7); Drug: bevacizumab (Avastin); Drug: irinotecan; Drug: Leucovorin; Drug: 5-FU
- UGT1A1 non-genotyping (Experimental): The investigators will maintain the dosage of irinotecan by 180mg/m2
  Interventions: Genetic: UGT1A1 non-genotyping; Drug: bevacizumab (Avastin); Drug: irinotecan; Drug: Leucovorin; Drug: 5-FU

INTERVENTIONS:
Genetic: UGT1A1 genotyping (6,6) — The investigators will use the regimen as following:
  Regimen for treatment consisted of bevacizumab (Avastin) 5mg/Kg (IV infusion) on day 1, follow by irinotecan (180 mg/m2 as a 120-min IV infusion), Leucovorin (400 mg/m2 IV infusion over 2 hours), and 5-FU (2800 mg/m2 IV infusion over a 46-hour period), repeated every 2 weeks.
  After 2 cycles of each different dose of irinotecan, we will observe the adverse effects (AEs) of hematological / non-hematological. If the grade is under the grade 2, we will escalate the dose of 30 mg/m2 gradually. The estimated maximal dose of irinotecan is 260 mg/m2.
  Other Names: UGT1A1*1*1
  Arms: UGT1A1 genotyping (6,6)
Genetic: UGTIA1 genotyping (6,7) — The investigators will use the regimen as following:
  Regimen for treatment consisted of bevacizumab (Avastin) 5mg/Kg (IV infusion) on day 1, follow by irinotecan (180 mg/m2 as a 120-min IV infusion), Leucovorin (400 mg/m2 IV infusion over 2 hours), and 5-FU (2800 mg/m2 IV infusion over a 46-hour period), repeated every 2 weeks.
  After 2 cycles of each different dose of irinotecan, we will observe the adverse effects (AEs) of hematological / non-hematological. If the grade is under the grade 2, we will escalate the dose of 30 mg/m2 gradually. The estimated maximal dose of irinotecan is 240 mg/m2.
  Other Names: UGT1A1*1*28
  Arms: UGTA1T1 genotyping (6,7)
Genetic: UGTIA1 genotyping (7,7) — The investigators will use the regimen as following:
  Regimen for treatment consisted of bevacizumab (Avastin) 5mg/Kg (IV infusion) on day 1, follow by irinotecan (120 mg/m2 as a 120-min IV infusion), Leucovorin (400 mg/m2 IV infusion over 2 hours), and 5-FU (2800 mg/m2 IV infusion over a 46-hour period), repeated every 2 weeks.
  After 2 cycles of each different dose of irinotecan, we will observe the adverse effects (AEs) of hematological / non-hematological. If the grade is under the grade 2, we will escalate the dose of 30 mg/m2 gradually. The estimated maximal dose of irinotecan is 180 mg/m2.
  Other Names: UGT1A1*28*28
  Arms: UGTA1T1 genotyping (7,7)
Genetic: UGT1A1 non-genotyping — The investigators will use the regimen as following:
  Regimen for treatment consisted of bevacizumab (Avastin) 5mg/Kg (IV infusion) on day 1, follow by irinotecan (180 mg/m2 as a 120-min IV infusion), Leucovorin (400 mg/m2 IV infusion over 2 hours), and 5-FU (2800 mg/m2 IV infusion over a 46-hour period), repeated every 2 weeks.
  Arms: UGT1A1 non-genotyping
Drug: bevacizumab (Avastin) — bevacizumab as target therapy
  Other Names: Avastin
Drug: irinotecan — irinotecan as escalating dose according to UGT1A1 genotyping
  Other Names: Campto
Drug: Leucovorin — combined with 5-FU
Drug: 5-FU — combined with irinotecan

SUMMARY:
Metastatic diseases were found in 20-25% of patients with initial diagnosis of colorectal cancer and developed in up to 50% of patients. Owing to limited post-treatment response of 5-fluorouracil (5-FU) combined with leucovorin (LV) obtained in mCRC (metastatic colorectal cancer) patients, other therapeutic agents with different mechanisms were considered, such as irinotecan, a potent inhibitor of topoisomerase I, which is involved in the unwinding of DNA during replication. Bevacizumab is a humanized monoclonal antibody that inhibits tumor angiogenesis by blocking vascular endothelial growth factor (VEGF) and was the first antiangiogenic agent approved for the treatment of cancer.

Infusional fluorouracil/leucovorin plus irinotecan-based regimen (FOLFIRI) with bevacizumab has been widely used as first-line treatment for patients with metastatic colorectal cancer (mCRC). Recently, the investigators have shown that prospective analysis of uridine diphosphate glucuronosyl transferase 1A1 (UGT1A1) genotyping for irinotecan dose escalation (FOLFIRI regimen) with combination of bevacizumab biweekly as the first-line setting in mCRC patients (ASCO Abstract #491 - 2013 Gastrointestinal Cancers Symposium).

In this study, the investigators will enroll approximately 320 mCRC patients (It was considered that an increase of response rate of 15% compared to conventional irinotecan dose of 180 mg/m2, and these were chosen as parameters with which to calculate the study power. Initial power calculation was suggested that a minimum of 140 patients in each group would be required to achieve statistical significance with a power of 80% at the 5% significance level. It is estimated that about 10% of 320 mCRC patients fail to complete the study). For these enrolled patients, the investigators will randomize and divide these patients into two groups: control group and study group. Control group includes mCRC patients who will receive the conventional regimen of FOLFIRI plus bevacizumab. Otherwise, patients in the study group will have genotyping of UGT1A1 before therapy, and dose escalating of irinotecan will depend on results of genotyping.

DETAILED DESCRIPTION:
Control group:

Regimen for treatment consisted of bevacizumab (Avastin) 5mg/Kg (IV infusion) on day 1, follow by irinotecan (180 mg/m2 as a 120-min IV infusion), LV (400 mg/m2 IV infusion over 2 hours), and 5-FU (2800 mg/m2 IV infusion over a 46-hour period), repeated every 2 weeks.

Study group: FOLFIRI (infusional fluorouracil/leucovorin plus irinotecan) + Bevacizumab. The dosage of irinotecan is adjusted to the UGT1A1 genotyping

The wild-type (6/6) of UGT1A1:

Regimen for treatment consisted of bevacizumab (Avastin) 5mg/Kg (IV infusion) on day 1, follow by irinotecan (180 mg/m2 as a 120-min IV infusion), LV (400 mg/m2 IV infusion over 2 hours), and 5-FU (2800 mg/m2 IV infusion over a 46-hour period), repeated every 2 weeks.

After 2 cycles of each different dose of irinotecan, we will observe the adverse effects (AEs) of hematological / non-hematological. If the grade is under the grade 2, we will escalate the dose of 30 mg/m2 gradually. The estimated maximal dose of irinotecan is 260 mg/m2.

The (6,7) type of UGT1A1:

Regimen for treatment consisted of bevacizumab (Avastin) 5mg/Kg (IV infusion) on day 1, follow by irinotecan (180 mg/m2 as a 120-min IV infusion), LV (400 mg/m2 IV infusion over 2 hours), and 5-FU (2800 mg/m2 IV infusion over a 46-hour period), repeated every 2 weeks.

After 2 cycles of each different dose of irinotecan, we will observe the adverse effects (AEs) of hematological / non-hematological. If the grade is under the grade 2, we will escalate the dose of 30 mg/m2 gradually. The estimated maximal dose of irinotecan is 240 mg/m2.

The (7,7) type of UGT1A1:

Regimen for treatment consisted of bevacizumab (Avastin) 5mg/Kg (IV infusion) on day 1, follow by irinotecan (120 mg/m2 as a 120-min IV infusion), LV (400 mg/m2 IV infusion over 2 hours), and 5-FU (2800 mg/m2 IV infusion over a 46-hour period), repeated every 2 weeks.

After 2 cycles of each different dose of irinotecan, we will observe the adverse effects (AEs) of hematological / non-hematological. If the grade is under the grade 2, we will escalate the dose of 30 mg/m2 gradually. The estimated maximal dose of irinotecan is 180 mg/m2.

ELIGIBILITY:
Inclusion Criteria:

1. 20 y/o ≦ Age ≦ 80y/o
2. Either metachronous or synchronous mCRC can be enrolled
3. Female patients need not ready to be pregnant or breastfeeding
4. No major underlying diseases (such as cardiovascular, cerebrovascular, malignant hypertension, kidney, liver and other major diseases)
5. mCRC be proven by pathologists or radiologists
6. Subjects are willing to sign an inform consent form

Exclusion Criteria:

* Patients who do not meet the including criteria or unwilling to participate

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2014-08-13 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | three to six months

SECONDARY OUTCOMES:
Objective response rates | three to six months
overall survival | three to six months

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ho Memorial Hospital, Kaohsiung Medical University:, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Tsai HL, Huang CW, Lin YW, Wang JH, Wu CC, Sung YC, Chen TL, Wang HM, Tang HC, Chen JB, Ke TW, Tsai CS, Huang HY, Wang JY. Determination of the UGT1A1 polymorphism as guidance for irinotecan dose escalation in metastatic colorectal cancer treated with first-line bevacizumab and FOLFIRI (PURE FIST). Eur J Cancer. 2020 Oct;138:19-29. doi: 10.1016/j.ejca.2020.05.031. Epub 2020 Aug 20. PMID 32829105
- [Derived] Yeh YS, Tsai HL, Huang CW, Wang JH, Lin YW, Tang HC, Sung YC, Wu CC, Lu CY, Wang JY. Prospective analysis of UGT1A1 promoter polymorphism for irinotecan dose escalation in metastatic colorectal cancer patients treated with bevacizumab plus FOLFIRI as the first-line setting: study protocol for a randomized controlled trial. Trials. 2016 Jan 25;17:46. doi: 10.1186/s13063-016-1153-3. PMID 26811156